CLINICAL TRIAL: NCT06426901
Title: Effects of Tan Tui Exercises on Strength and Performance of Football Players.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/01835 Naveed Ullah
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Football Players
Keywords: Agility; Quickness; Change direction; Skills; Strength

STUDY DESIGN:
Intervention Model Description: group1 ,experimental group group 2 control group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: the group A will be received Tan Tui exercies (Experimental): Experimental Group A Springing Leg Forms." var-arranged sequences of movements that incorporate kicks, strikes, and blocks.
  Pattern Drills: Pattern drills involve repeating specific combinations of kicks, strikes, and blocks in a repetitive manner.
  Basic Kicking Drills: which involve ious types of kicks such as front kicks, sidekicks, roundhouse kicks, and crescent kicks.
  Stance Work: Practitioners work on a variety of stances, including horse stance (ma bu), bow stance (gong bu), and cat stance (mao bu).
  Forms (Taolu): These forms consist of predrills enhance muscle memory and the ability to execute techniques quickly and accurately.
  Conditioning: includes rigorous conditioning exercises to strengthen the legs and develop endurance.
  Sparring (San Shou):
  bouncing leg exercise intervention cycle lasted 6 weeks, 3 times a week for 30 minutes each. The intervention was split into two parts: motor learning in the first week and motor improvement in the last five weeks.
  .
  Interventions: Other: Effects of Tan Tui Exercises on Strength and Performance of Football Players.
- Controlled (No Intervention): Conventional exercises Squats: Squats are a foundational lower-body exercise that targets the quadriceps, hamstrings, glutes, and lower back.
  Bench Press: The bench press is a classic upper-body exercise that targets the chest, shoulders, and triceps.
  Power Cleans: Similar to the clean and jerk, power cleans are used to develop explosive power, especially in the legs and hips.
  Pull-Ups/Chin-Ups: Pull-ups and chin-ups strengthen the muscles of the upper back, shoulders, and arms.
  Push-Ups: Push-ups are a versatile exercise that works the chest, shoulders, triceps, and core.
  Lunges: Lunges are excellent for targeting the quadriceps, hamstrings, and glutes while also improving balance and stability.
  Core Exercises: Core strength is vital for stability and balance in football. Exercises like planks, Russian twists, and medicine ball throws target the core muscles.

INTERVENTIONS:
Other: Effects of Tan Tui Exercises on Strength and Performance of Football Players. — Tan Tui, Exercises Tan Tui, is a style of traditional Chinese martial art that emphasizes leg techniques, agility, and conditioning. Basic Kicking Drills. Stance Work. Forms (Taolu) Pattern Drills. Conditioning.Sparring (San Shou). This protocol will be implemented by District Physiotherapist who will visit the mentioned Football academies in group session.
  Arms: Experimental Group: the group A will be received Tan Tui exercies

SUMMARY:
Randomized controlled trial (RCT) to investigate the effects of Tan Tui exercises on the strength and performance of football players. Tan Tui can provide football players with a well-rounded approach to physical and mental development, which can contribute to enhanced performance, injury prevention, and personal improvement both on and off the field there is limited study available on the effectiveness of Tan Tui exercises.

DETAILED DESCRIPTION:
Tan Tui training develops mental fortitude, focus, and discipline. Football players can benefit from better concentration, emotional resilience, and the capacity to remain calm under pressure. While football generally focuses on offensive and defensive strategies, mastering Tan Tui self-defense techniques can teach players with real abilities for personal protection off the field. Tan Tui can help with injury prevention by increasing flexibility and body awareness. Tan Tui practitioners are frequently more equipped to avoid strains and sprains. The meditative aspects of Tan Tui training can help football players manage stress and anxiety, improving their mental well-being and overall quality of life.

ELIGIBILITY:
Inclusion Criteria Male Player

* Player of academy from last 1 year
* Aged 18-35 years.
* BMI (19-29)

Exclusion Criteria:

* • Surgical History

  * Fracture History
  * Meniscal pathology
  * Knee injury due to trauma

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Hand Held Dynamometer | 6 weeks
  Modified Hand Held Dynamometers (will assess the power of lower limb Muscle)

SECONDARY OUTCOMES:
Agility T-Test | 6th week
  The Agility T-Test is a fitness test that is commonly used in sports and physical fitness training to assess an individual's agility, speed, and quickness. It is especially common in sports requiring quick changes of direction, such as basketball, soccer, football, and tennis. The exam is named after the T-shaped running course that participants must complete in the shortest amount of time.

CONTACTS AND LOCATIONS:
Overall Officials: Riafat Mehmood, Principal Investigator — Riphah International University
Locations (1):
- Timergara Football club, Dīr, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No